CLINICAL TRIAL: NCT00179257
Title: The Effectiveness of Sertraline in Patients Who Have Had Inadequate Response to
Brief Title: The Effectiveness of Sertraline in Patients Who Have Had Inadequate Response to Escitalopram
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Richard C. Shelton, Director of Mood Disorders Clinic, Vanderbilt University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lexapro Failure Study
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-06

CONDITIONS: Major Depressive Disorder
Keywords: Failure to Escitalopram
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Sertraline

INTERVENTIONS:
Drug: sertraline (Zoloft)

SUMMARY:
The purpose of this is to determine the efficacy, safety, and tolerability of sertraline in patients with major depressive disorder (MDD) who have shown inadequate response ot escitalopram.

DETAILED DESCRIPTION:
Eight week open-label flexible dose trial in adult outpatients diagnosed with Major Depressive Disorder (MDD) who have had a prior failure with escitalopram. Failure is operationally defined as either premature discontinuation because of side effects or the report of an incomplete response to escitalopram, minimum dose 10mg/day, maintain for 3 weeks or more. 10mg/day was chosen because 1) it is the most commonly prescribed single dose of escitalopram in clinical practice, 2) it is equivalent to approx. 30mg/day of arcemic citalopram and 3) escitalopram has very high potency at the serotonin transporter (Ki=1.1); this means that escitalopram would be expected to saturate the transporter at relatively low doses. A total of twenty patients will be treated.

ELIGIBILITY:
Inclusion Criteria:

* Primary DSM-IV diagnosis of Major Depressive episode of MDD without psychotic symptoms. Additional axis I diagnoses will be permitted only if they are identified as secondary diagnoses
* Ham-D 21 item score of greater than or equal to 18
* Age 18 and above
* Ability and willingness to provide consent for participation
* Failure to respond to escitalopram

Exclusion Criteria:

* Diagnosis of Bipolar Disorder or any psychotic disorder
* Alcohol or drug abuse or dependence currently or in the last 6 months
* A history of non-response or intolerance to sertraline at least 50 mg. for at least 4 weeks or more
* Concomitant use of another antidepressant or use of an antidepressant within 2 weeks of baseline (4 weeks for fluoxetine)
* Use within 1 week of baseline, or concomitant use of any psychotropics with the exception of zolpidem for sleep
* Use within 4 weeks of baseline or concomitant use of benzodiazepines with the exception of PRN use of diazepam 10 mg/day or its equivalent
* Presence of serious and/or unstable medical condition
* Score of 3 or 4 on the suicide item (item 3) of the Ham-D scale
* Known sensitivity of sertraline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2004-06; Study Completion 2005-03

PRIMARY OUTCOMES:
Quality of Life, Enjoyment, and Satisfaction Scale (Q-LES-Q)
Hamilton Rating Scale for Depression (21-item) total score
Clinical Global Impressions - Improvement Scale

SECONDARY OUTCOMES:
Hamilton Anxiety Scale Total score
Clinical Global Impressions - Severity Scale

CONTACTS AND LOCATIONS:
Overall Officials: Richard C Shelton, MD, Principal Investigator — Vanderbilt University Medical Center